CLINICAL TRIAL: NCT00419692
Title: An Open Label, Repeat Dose, Dose Escalation Study Conducted in RLS Patients to Characterize Pharmacokinetics and Food Effect of Ropinirole Controlled Release for RLS
Brief Title: Restless Legs Patient Study On Absorption, Distribution, Metabolism And Excretion Of Ropinirole And The Effect Of Food
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ROR106470
Record Dates: First submitted 2007-01-05; First posted 2007-01-09 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Restless Legs Syndrome
Keywords: pharmacokinetic,; RLS; formulation,; food effect,; controlled release for RLS,; SK&F101468,
MeSH Terms: conditions — Restless Legs Syndrome | interventions — ropinirole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Sequence WAXBYZCDE (Experimental): Subjects will receive ropinirole as follows W: 1 x 0.5 mg CR-RLS (normal fed), A: 1 x 1 mg CR-RLS (fasted), X: 1 x 2 mg CR-RLS (normal fed), B: 1 x 3 mg CR-RLS (fasted), Y: 2 x 2 mg CR-RLS (normal fed), Z: (2 x 2 mg) + (1 x 1 mg) CR-RLS (normal fed), C: 1 x 6 mg CR-RLS (fasted), D: 1 x 6 mg CR-RLS (high fat fed) and E: 2 x 3 mg CR-RLS (fasted).
  Interventions: Drug: Ropinirole
- Sequence WAXBYZCED (Experimental): Subjects will receive ropinirole as follows W: 1 x 0.5 mg CR-RLS (normal fed), A: 1 x 1 mg CR-RLS (fasted), X: 1 x 2 mg CR-RLS (normal fed), B: 1 x 3 mg CR-RLS (fasted), Y: 2 x 2 mg CR-RLS (normal fed), Z: (2 x 2 mg) + (1 x 1 mg) CR-RLS (normal fed), C: 1 x 6 mg CR-RLS (fasted), E: 2 x 3 mg CR-RLS (fasted) and D: 1 x 6 mg CR-RLS (high fat fed).
  Interventions: Drug: Ropinirole
- Sequence WAXBYZDCE (Experimental): Subjects will receive ropinirole as follows W: 1 x 0.5 mg CR-RLS (normal fed), A: 1 x 1 mg CR-RLS (fasted), X: 1 x 2 mg CR-RLS (normal fed), B: 1 x 3 mg CR-RLS (fasted), Y: 2 x 2 mg CR-RLS (normal fed), Z: (2 x 2 mg) + (1 x 1 mg) CR-RLS (normal fed), D: 1 x 6 mg CR-RLS (high fat fed), C: 1 x 6 mg CR-RLS (fasted) and E: 2 x 3 mg CR-RLS (fasted).
  Interventions: Drug: Ropinirole
- Sequence WAXBYZDEC (Experimental): Subjects will receive ropinirole as follows W: 1 x 0.5 mg CR-RLS (normal fed), A: 1 x 1 mg CR-RLS (fasted), X: 1 x 2 mg CR-RLS (normal fed), B: 1 x 3 mg CR-RLS (fasted), Y: 2 x 2 mg CR-RLS (normal fed), Z: (2 x 2 mg) + (1 x 1 mg) CR-RLS (normal fed), D: 1 x 6 mg CR-RLS (high fat fed), E: 2 x 3 mg CR-RLS (fasted) and C: 1 x 6 mg CR-RLS (fasted).
  Interventions: Drug: Ropinirole
- Sequence WAXBYZECD (Experimental): Subjects will receive ropinirole as follows W: 1 x 0.5 mg CR-RLS (normal fed), A: 1 x 1 mg CR-RLS (fasted), X: 1 x 2 mg CR-RLS (normal fed), B: 1 x 3 mg CR-RLS (fasted), Y: 2 x 2 mg CR-RLS (normal fed), Z: (2 x 2 mg) + (1 x 1 mg) CR-RLS (normal fed), E: 2 x 3 mg CR-RLS (fasted),C: 1 x 6 mg CR-RLS (fasted) and D: 1 x 6 mg CR-RLS (high fat fed).
  Interventions: Drug: Ropinirole
- Sequence WAXBYZEDC (Experimental): Subjects will receive ropinirole as follows W: 1 x 0.5 mg CR-RLS (normal fed), A: 1 x 1 mg CR-RLS (fasted), X: 1 x 2 mg CR-RLS (normal fed), B: 1 x 3 mg CR-RLS (fasted), Y: 2 x 2 mg CR-RLS (normal fed), Z: (2 x 2 mg) + (1 x 1 mg) CR-RLS (normal fed), E: 2 x 3 mg CR-RLS (fasted), D: 1 x 6 mg CR-RLS (high fat fed) and C: 1 x 6 mg CR-RLS (fasted).
  Interventions: Drug: Ropinirole

INTERVENTIONS:
Drug: Ropinirole — Subjects will receive ropinirole 0.5 mg for first 7 days, 1 mg from Day 8-14, 2 mg from Day 15-21, 3 mg from Day 22-28, 4 mg from Day 29-35, 5 mg from Day 36-42 and 6 mg from Day 43-51.

SUMMARY:
This study in RLS patients is designed to assess the affect food has on the absorption, distribution, metabolism and excretion of ropinirole (by dosing some patients in the fasted state and other patients following a high-fat breakfast), and to assess the difference in absorption, distribution, metabolism and excretion of ropinirole if patients are given two 3mg ropinirole tablets versus one 6mg tablet.

ELIGIBILITY:
Inclusion criteria:

* Patients with a diagnosis of RLS
* Body mass index of 18 to 32 kg/m², with a body weight of at least 50 kg
* Normal blood pressure pre-study
* Light smokers only (<20/day)

Exclusion criteria:

* History of postural hypotension or faints
* Secondary RLS
* Patients who suffer from a primary sleep disorder other than RLS
* Patients diagnosed with movement disorders
* Patients with unstable medical conditions
* Patients with personal or family history of adverse reactions or hypersensitivity to the study drug
* Patients with abnormal laboratory values
* Patients with hepatitis or HIV
* Patients who abuse alcohol or drugs
* Patients taking the following medications: dopamine agonists (including ropinirole), dopamine antagonists (e.g., metoclopramide and domperidone), levodopa/carbidopa

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2006-08-24 (Actual); Primary Completion 2006-12-12 (Actual); Study Completion 2006-12-12 (Actual)

PRIMARY OUTCOMES:
Ropinirole AUC (area under the plasma concentration-time curve) over the dosing interval Ropinirole maximum plasma concentration | dosing interval

SECONDARY OUTCOMES:
Time to attain the maximum plasma concentration Time taken for ropinirole concentration to fall to half initial value Incidence of adverse events Vital signs, ECG and clinical laboratory data As above, but for ropinirole metabolites | Time taken for ropinirole concentration to fall to half initial value

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- GSK Investigational Site, Berlin, Germany
- GSK Investigational Site, George, South Africa

REFERENCES:
- See also: Results for study ROR106470 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/ROR106470?search=study&search_terms=ROR106470#rs